CLINICAL TRIAL: NCT01712477
Title: Propofol Versus Midazolam for Sedation in Mechanically Ventilated Critically Ill Patients Who Presented With Traumatic Brain Injury: Cytokine Response and Neuropsychological Assessment (IRRC#1201M)
Brief Title: A Comparison of Propofol Versus Midazolam to Sedate Critically Brain Injury; Measurement of Cytokine Response and Assessment of Function
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruiting
Sponsor: Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: r039226; IRRC#1201M (Other: Michigan State University IRB)
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2025-06-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous sedation with propofol (Active Comparator): Traumatic brain injured patient, already requiring sedation. Intervention is sedation with intravenous propofol during mechanical ventilation
  Interventions: Drug: Intravenous sedation using propofol
- Intravenous sedation with midazolam (Active Comparator): Patients with traumatic brain injury requiring mechinical ventilation. Intervention is intravenous midazolam for sedation at variable doses to achieve adequite sedation levels
  Interventions: Drug: Intravenous sedation with midazolam

INTERVENTIONS:
Drug: Intravenous sedation using propofol — Patients will be given intravenous sedation for treatment of traumatic brain injury requiring mechanical ventilation
  Arms: Intravenous sedation with propofol
Drug: Intravenous sedation with midazolam — patients with severe traumatic brain injury requiring mechanical ventilation and sedation will be sedated with midazolam
  Other Names: Versed
  Arms: Intravenous sedation with midazolam

SUMMARY:
This is a prospective randomized controlled pilot study in traumatic brain injury (TBI) patients who are sedated with either propofol or midazolam to compare the cytokine response and neuropsychological outcomes with and without elevated blood alcohol levels.

Sedation is part of the standard treatment in patients with a TBI and has been proposed as a neuroprotective intervention in head-injured patients. Sedative regimens, such as midazolam and propofol, are not standardized and it is unclear whether sedation has a significant impact on recovery and outcome. A review of propofol versus midazolam in mechanically ventilated patients shows evidence that both provide effective sedation but there is lack of data to support one sedative over the other.

Cytokines are released in response to tissue injury and act to generate a variety of physiologic responses. The cytokine elevation has been correlated with the extent of tissue injury. This study will compare the cytokine distribution patterns at specific posttraumatic time points in patients with a TBI sedated with either propofol or midazolam. Additional analysis will compare the cytokine response in patients whom had elevated blood alcohol levels with those with normal levels. Neuropsychological testing will also be performed to determine the extent of brain injury and recovery.

DETAILED DESCRIPTION:
The purpose of this research is to compare the effectiveness, length of time from cessation of sedation till extubation, recovery time, duration of admission to the ICU, recovery of brain function, cytokine response, and complication rate of propofol versus midazolam when used for sedation in patients with traumatic brain injury (TBI) with or without elevated blood alcohol levels. Since this type of trauma patient will require significant medical care upon admission to the emergency room (ER) and the family will be concerned about the injuries, the patient and/or family will not be approached about the research study during this time. At the earliest possible time following neurointensive (NICU) or intensive care (ICU) admission, an informed consent will be obtained from the patient. Depending on the severity of the head injury, the patients may not be able to sign an informed consent. In this case, the consent will be obtained from next-of-kin or a legal guardian. No interventions or study research will be conducted on the patient until the consent is obtained.

Standard blood panels are drawn for every trauma patient regardless of whether or not the patient is a participant of the research protocol, including blood alcohol levels. During the trauma workup in ER, it is standard of care to draw an extra vial in case additional lab tests are needed. After consent is obtained, the research team will obtain the extra vial from the Sparrow Lab to perform cytokine and blood cell phenotype measurements for the research study. Typically 0.5-1.0 ml of whole blood is needed for these measurements and that can be taken from the standardized EDTA tube that is drawn on admission. This small amount of blood sample would otherwise be discarded. Plasma cytokines and cell phenobype IL-1, IL-3, IL-6, IL-8, IL-10, IL-17, TNF-¦Á, TGF-¦Â, G-CSF, GM-CSF, SCF, FGF, and IGF-II will be performed by Luminex-based mutiplex assay and ELISA. In addition to the ER analysis, left over blood will be used from the EDTA tubes at 24 hours, day 3 and day 7 after admission. These additional measurements will be taken from the routine morning laboratory blood draws which are done on all intubated patients to evaluate electrolytes. No additional blood will be drawn for the research and the study will only be using left over blood already drawn for standard of care labs that are done on all intubated patients.

Once consented, the patients will be randomized to treatment group by random allocation process using Research Randomizer (Urbaniak, G. C., & Plous, S. Version 3.0 Computer software]. The patient and family will be blinded to which sedation is given. Nurses and physicians will not be blinded as they will be administering the sedatives. Although the patients will receive randomized sedation, these patients would be administered either propofol or midazolam even if they were not included in this research. The only modification for research purposes is the randomization of sedation medication by the randomizer rather than the physician. Currently, the providers in the research team do not have a preference of one type of sedation medication over the other.

Once randomized, patients allocated to the propofol group will be initiated with a 0.5-1 mg/kg i.v. bolus followed by repeated 10-20 mg doses at variable intervals (approximately 15 s, at the discretion of the physician/nurse) until an appropriate level of sedation will be achieved (NICU protocol), which will be subsequently titrated to achieve a target Richmond Agitation-Sedation Scale (+4 = combative to -5 = unarousable) (Sessler et al. The Richmond Agitation-Sedation Scale.Am J Respir Crit Care Med 2002; 166:1338-1344). Nurses will note pre-sedation levels based on the Richmond Agitation-Sedation Scale. While undergoing sedation, target sedation will be defined when the Richmond Agitation-Sedation Scale meets a score of -4 to -5. Patients randomized to the midazolam group will be initiated with 0.5-1.0 mg with incremental dosing at intervals of approximately 1-3 min until a level of sedation will be achieved at a target Richmond Agitation-Sedation scale sedation score (per NICU protocol).

Management of all trauma patients include a careful history taking for alcoholism with referral for further evaluation or treatment when indicated, and determination whether other drugs are also being used. All patients with an elevated alcohol level require a medical social service consultation and all patients with a TBI require a neuropsychology consultation, both consultations are standard of care. The neuropsychological testing conducted after extubation is also standard of care. The neuropsychological evaluations will be measured based on the following assessments: intellectual functioning, language processing, visuospatial processing, attention, concentration, verbal learning, memory, executive functioning, sensory, perception, motor, strength, and personal assessment. The level of impairment will be based on a scale from zero to seven. Data will be collected until the patient is discharged from the hospital. The clinical records from the neuropsychologist will be reviewed to analyze the progression of the patient's outcome. Similar to all trauma patients, the patients enrolled in this study will be offered continued care with neuropsychology as well as the option to withdrawal all care if competent to make independent decisions.

Throughout the study consciousness will be measured using the Glasgow Coma Score (GCS) from the time of presentation to the ER and two times each day until the patient is discharged from the NICU or ICU (routinely done on TBI patients). The Injury severity scores (ISS) will be recorded from admission (done on all trauma patients). Recovery of consciousness will be determined by measurement of the acute physiology and chronic health evaluation (APACHE) III modification of the Glasgow coma score to allow for scoring of the verbal component in intubated patients. Patients will be judged to be awake when the Glasgow coma score was > or = 12.

The following will be recorded from the Sparrow medical record for each patient: gender, age, sex, weight, primary diagnosis, significant co morbidities, blood alcohol level at admission, intracranial pressure measurements (standard of care for TBI patients), time of starting and finishing of the sedation, total amount of medications given, any restraint required, additional oxygen required, resuscitative measures required, time of transfer out of the unit, and time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 Years or older
* Males or Females
* Primary diagnosis of TBI, subarachnoid hemmorhage (SAH), intracranial hemmorhage (ICH), stroke
* Requires mechanical ventilation
* Requires or is receiving continuous IV sedation

Exclusion Criteria:

* Glascow Coma Score (GCS) of 3 persisting from the scene with bilaterally fixed dilated pupils with no appreciable chance of survival
* The inability to identify a next of kin or guardian to give consent if patient unable to consent
* Pregnant
* Allergy or contraindication to propofol
* Allergy to contraindication to midalozam
* Status epilepticus
* Current neuromuscular blockade
* Patient with a known hypersensitivity to propofol or midalozam
* Allergies to eggs, egg products, soybeans or soy products
* Acute narrow-angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chet A Morrison, M.D., Principal Investigator — Michigan State University
Locations (1):
- Sparrow Health System, Lansing, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Sedation With Propofol
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous Sedation With Propofol
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychologic Outcome
Description: Extent of functional deficits from underlying traumatic brain injury
Time Frame: 30 days
Population: Only one participant was enrolled and data analysis was not completed
Groups:
- Intravenous Sedation With Propofol: Traumatic brain injured patient, already requiring sedation. Intervention is sedation with intravenous propofol during mechanical ventilation
  Intravenous sedation using propofol: Patients will be given intravenous sedation for treatment of traumatic brain injury requiring mechanical ventilation
  Outcome measure: Survival and transfer to neurocognitive rehabilitation
Arm/Group | Intravenous Sedation With Propofol
Number analyzed (Participants) | 0

2. Secondary Outcome: Cytokine Levels Correlating to Extent of Injury
Description: cytokine levels will be measured to see if there is meaningful correlation between groups.
  unable to correlate due to closure of study
Time Frame: 30 days
Population: Only one participant was enrolled and data analysis was not completed.
Arm/Group | Intravenous Sedation With Propofol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Protocol closed due to low enrollment
Groups:
- Intravenous Sedation With Propofol: Traumatic brain injured patient, already requiring sedation. Intervention is sedation with intravenous propofol during mechanical ventilation
  Intravenous sedation using propofol: Patients will be given intravenous sedation for treatment of traumatic brain injury requiring mechanical ventilation
  Outcome measure: Survival and transfer to neurocognitive rehabilitation.
  No adverse events noted
Arm/Group | Intravenous Sedation With Propofol
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes